CLINICAL TRIAL: NCT02711371
Title: Long-term Effects of Cannabis Use on Social and Emotional Brain Processes in Dependent Cannabis Users After a 28 Day Abstinence Period
Brief Title: Social and Emotional Brain Function in Cannabis Users
Status: Completed | Type: Observational
Sponsor: University of Electronic Science and Technology of China (Other)
Collaborators: German Research Foundation (Other); University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Prof. Dr. rer. nat., University of Electronic Science and Technology of China
Other Study IDs: ART_Can_01
Record Dates: First submitted 2016-03-04; First posted 2016-03-17 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Cannabis Dependence
Keywords: addiction; cannabis; fMRI
MeSH Terms: conditions — Marijuana Abuse; Behavior, Addictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cannabis Dependence: Cannabis dependent individuals according to DSM 4 criteria, aged 18-40 years
  Interventions: Other: fMRI
- Healthy: Healthy controls, socio-demographically matched
  Interventions: Other: fMRI

INTERVENTIONS:
Other: fMRI

SUMMARY:
The aim of this functional magnetic resonance imaging (fMRI) study is to find out whether and how social and emotional brain function are altered in dependent cannabis users relative to healthy non-using control subjects after a 28 supervised abstinence period. Previous research in cannabis users has predominantly focused on cognitive functions. Moreover, studies have implicated that observed deficits in cannabis users may regenerate after a prolonged abstinence period. Findings might provide important information with respect to relapse vulnerability.

ELIGIBILITY:
Inclusion Criteria:

* Cannabis dependence according to DSM 4 criteria
* 28 days of supervised abstinence

Exclusion Criteria:

* other DSM 4 diagnosis
* neurological disorders

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cannabis dependent individuals
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
fMRI neural activation patterns of social-emotional brain processes after 28 day abstinence | one timepoint = fMRI assessment after 28 day abstinence period
  Activity patterns in core regions of the emotion processing & addiction-related brain networks (e.g. striatal regions, insular cortex, prefrontal cortex) will be assessed after 28-days of abstinence. Alterations will be determined by comparison with matched non-drug using controls

SECONDARY OUTCOMES:
Ratings of subjective experience (pleasantness, rewarding value) will be assessed after 28 days of abstinence | one timepoint = during fMRI assessment after 28 day abstinence period
  Self-reported ratings of pleasantness & rewarding value during soft-pleasant touch.
Relapse interview assessed with Timeline-Followback Method | one timepoint = 24 months post-fMRI-session
  Association between fMRI neural correlates and drug use during follow up period as predictor of relapse

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bonn / Department of Psychiatry, Bonn, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Zimmermann K, Yao S, Heinz M, Zhou F, Dau W, Banger M, Weber B, Hurlemann R, Becker B. Altered orbitofrontal activity and dorsal striatal connectivity during emotion processing in dependent marijuana users after 28 days of abstinence. Psychopharmacology (Berl). 2018 Mar;235(3):849-859. doi: 10.1007/s00213-017-4803-6. Epub 2017 Dec 2. PMID 29197984